CLINICAL TRIAL: NCT00821782
Title: A Randomized, Open-Label Study Comparing Levofloxacin Once-Daily 750 mg PO for 5 Days and Azithromycin Once-Daily 500 mg on Day One and Then 250 mg Days 2 Through 5 In a Microbiologic Evaluation for Emergence of Resistance in the Oropharyngeal Flora of Healthy Subjects
Brief Title: Evaluation of Bacteria in the Mouth and Throat of Healthy Adults Before and After the Administration of Either Levofloxacin or Azithromycin, Both Antibiotic Medications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012235
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Healthy Volunteer
Keywords: Bacteria; Oral flora bacteria; Resistance
MeSH Terms: interventions — Levofloxacin; Azithromycin

INTERVENTIONS:
Drug: Levofloxacin; Azithromycin

SUMMARY:
Evaluation of bacteria in the mouth and throat before study drug ( Levofloxacin, floroquinolone antibiotic and Azithromycin, a macrolide antibiotic) is started and then periodically for 6 weeks after the last dose of study drug is taken

DETAILED DESCRIPTION:
This is a randomized, open-label, single center, exploratory, Phase 1 study to explore changes and resistance patterns of bacteria in the oral flora of healthy male and female adult subjects. The study is to enroll approximately 140 healthy subjects. Approximately 70 subjects are to receive levofloxacin once daily for 5 days and 70 are to receive azithromycin once daily for 5 days. Male or female healthy subjects, 18 years or older may participate. Subjects will be treated on an outpatient basis at a Phase 1 facility. Laboratory testing (blood and urine collection) and microbiologic testing (throat swab) will be performed before dosing with study drug at the Study Entry (Visit 1). Subjects will return daily to the testing facility for their once-daily dosing of study drug for Visits 2 through 5 for a total of 5 consecutive days. At Visit 5 laboratory and microbiologic testing will be performed. Subjects will again return to the testing facility for the 2-Week (Visit 6), 4-Week (Visit 7) and 6-Week (Visit 8) Post-Therapy Visits to undergo microbiologic testing (throat swab). The primary endpoint is the emergence of bacterial resistance in the oropharyngeal flora starting prior to the initiation of study drug through a 6-week observation period. Microbiologic testing (throat swab) will be conducted prior to dosing on Day 1 and following dosing on Days 5, 19, 33, and 47. Safety assessments will be conducted prior to drug administration, during study drug treatment, and at the end-of-therapy visit. These included clinical laboratory evaluations, vital signs, physical examinations, pregnancy testing, and collection of adverse events. Serious adverse events will be collected for 30 days following the last dose of study drug. Levofloxacin Once-Daily 750 mg PO For 5 Days And Azithromycin Once-Daily 500 mg PO On Day One And Then 250 mg On Days 2 Through 5

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Healthy on the basis of a pre-study physical examination, medical history, and the laboratory results of blood hematology, biochemistry, and urinalysis performed within 24 hours before the first dose
* Renal function tests must be within the normal laboratory reference ranges
* Normotensive with sitting (5 minutes) blood pressure between the range of 90 to 140 mmHg systolic, inclusive, and 50-90 mmHg diastolic, inclusive
* Normal temperature for at least 72 hours. Normal defined as >36.0 C (96.8 F) to <37.5 C (99.5 F)
* Weight as defined by BMI range of 18 to 32 kg/m2, inclusive
* Must have read and signed the informed consent document before the first study-related procedure indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* History of allergy or serious adverse reaction to levofloxacin or any other quinolone or to azithromycin or any other macrolide
* Clinically significant abnormal laboratory values
* Previous systemic antimicrobial therapy within 3 months of Study Entry for any reason
* Hospitalized for any cause within 3 months prior to Study Entry
* Current drug abuse, alcohol abuse, or homelessness
* Requirement for any prescription or non-prescription medication or supplements such as vitamins and herbal supplements, except for paracetamol (acetaminophen) for the treatment of headache and other pain, hormone replacement therapy, and birth control medication upon study entry and during study conduct
* Pregnancy or breastfeeding
* Has received an experimental drug or medical device within the previous 3 months or involvement in any other experimental protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2006-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the emergence or worsening of bacterial resistance in the mouth and throat through six weeks after completion of the antibiotic

SECONDARY OUTCOMES:
All bacterial species cultured from the mouth and throat will be recorded. Each bacterial species seen at baseline, the proportion of subjects in which there was bacterial resistance will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC

REFERENCES:
- [Derived] Nord CE, Peterson J, Ambruzs M, Fisher AC. Levofloxacin versus azithromycin on the oropharyngeal carriage and selection of antibacterial- resistant streptococci in the microflora of healthy adults. Curr Med Res Opin. 2009 Jun;25(6):1461-7. doi: 10.1185/03007990902953468. PMID 19419343
- See also: N OPEN-LABEL RANDOMIZED STUDY COMPARING LEVOFLOXACIN 750 MG/DAY FOR 5 DAYS AND AZITHROMYCIN 500 MG ON DAY 1 AND 250MG ON DAYS 2-5 IN A MICROBIOLOGIC EVALUATION FOR EMERGENCE OF BACTERIAL RESISTANCE IN HEALTHY SUBJECTS' OROPHARYNGEAL FLORA — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=936&filename=CR012235_CSR.pdf